CLINICAL TRIAL: NCT03739268
Title: GLP-1-mediated Gluco-metabolic Effects of Bile Acid Sequestration
Acronym: SeveX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SeveX2018
Record Dates: First submitted 2018-10-11; First posted 2018-11-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: bile acid
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sevelamer (Active Comparator): Patients with type 2 diabetes treated with sevelamer
  Interventions: Drug: Sevelamer
- placebo (Placebo Comparator): Patients with type 2 diabetes treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sevelamer — Sevelamer powder dissolved in water 1,600 mg three times a day for 17 days
  Other Names: Renvela
  Arms: sevelamer
Drug: Placebo — placebo powder dissolved in water 1,600 mg three times a day for 17 days
  Arms: placebo

SUMMARY:
The objective of this study is to investigate the potential GLP-1-mediated contribution to the well-established glucose-lowering effect of sevelamer-induced bile acid sequestration . Exendin9-39 has been demonstrated to act as a potent and specific GLP-1 receptor antagonist with no partial agonistic potential and is considered a useful tool in the assessment of GLP-1 physiology. The aim is to evaluate any contribution of sevelamer-induced GLP-1 secretion to the reduced plasma glucose concentrations observed after treatment with sevelamer. A randomised placebo-controlled cross-over study involving two 17-day treatment periods with sevelamer and placebo, respectively, in metformin-treated patients with type 2 diabetes, will be conducted. The impact of bile acid sequestration on GLP-1 secretion and effect will be examined during two randomised experimental days after 15 and 17 days of treatment with sevelamer (1,600 mg three times a day) and placebo, respectively. During each of these two experimental days, a meal test with concomitant exendin9-39 infusion or placebo will be performed (for evaluation of any GLP-1-mediated effects). Postprandial plasma glucose excursion is the primary endpoint, and secondary endpoints include postprandial plasma/serum excursions of insulin, C-peptide, GLP-1, glucagon, glucose-dependent insulinotropic polypeptide (GIP), glucagon-like peptide-2 (GLP-2), peptide YY (PYY), oxyntomodulin, ghrelin, fibroblast growth factor (FGF)-19, FGF-21, C4 (an intermediate in the de novo synthesis of bile acids), cholecystokinin (CCK), bile acids and plasma lipids. Furthermore, gastric emptying, gallbladder emptying, liver fat content, appetite and ad libitum food intake will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 3 months (diagnosed according to the criteria of the World Health Organization (WHO))
* Men and postmenopausal women
* Metformin applied as the only glucose-lowering drug
* Caucasian ethnicity
* Normal haemoglobin
* Age above 40 years and below 75 years
* BMI >23 kg/m2 and <35 kg/m2
* Informed and written consent

Exclusion Criteria:

* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* Nephropathy (serum creatinine >150 µM and/or albuminuria)
* Hypo- or hyperthyroidism
* Hypo- or hypercalcaemia
* Hypo- or hyperphosphataemia
* Active or recent malignant disease
* Treatment with medicine that cannot be paused for 12 hours
* Treatment with oral anticoagulants
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Any condition considered incompatible with participation by the investigators

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
plasma glucose | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Postprandial plasma glucose (PG) excursion (AUC240 min)

SECONDARY OUTCOMES:
Postprandial responses of glucagon-like peptide-1 (GLP-1) | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of GLP-1
Postprandial responses of glucose-dependent insulinotropic polypeptide (GIP) | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of glucose-dependent insulinotropic polypeptide (GIP)
Postprandial responses of glucagon-like peptide-2 (GLP-2) | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of glucagon-like peptide-2 (GLP-2)
Postprandial responses of Glucagon | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of Glucagon
Postprandial responses of peptide YY (PYY) | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of peptide YY (PYY)
Postprandial responses of Insulin and c-peptide | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of Insulin and c-peptide as a insulin/c-peptide ratio
Postprandial responses of Ghrelin | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of Ghrelin
Postprandial responses of fibroblast growth factor (FGF)-19 | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of fibroblast growth factor (FGF)-19
Postprandial responses of fibroblast growth factor (FGF)-21 | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of fibroblast growth factor (FGF)-21
Postprandial responses of Bile acids | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of Bile acids
Postprandial responses of cholecystokinin (CCK) | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of cholecystokinin (CCK)
Postprandial responses of plasma lipids | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of plasma lipids
Postprandial responses of Amino acids | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Meal response of Amino acids
Gastric emptying | -30 minutes to 240 minutes with ingestion of a meal and paracetamol at 0 minutes
  Gastric emptying measured by paracetamol absorption test. Paracetamol is ingested along with meal, the appearance in blood will be calculated as a measure of gastric emptying.
Rate of gall bladder emptying | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  Gall bladder volumen measured by ultrasound over time after a meal (see time frame below). The rate of gall bladder emptying will be calculated
Liver stiffness and fat | At initiation and after 15 days of treatment with sevelamer/placebo
  Liver stiffness and fat content measured by fibroscan
Appetite measured by visual analog scale | -30 minutes to 240 minutes with ingestion of a meal at 0 minutes
  We assessed appetite parameters (hunger, satiety, fullness, prospective food consumption) and well-being, nausea, and thirst by visual analogue scales. Overall appetite score (OAS) will be calculated as (satiety + fullness + (100 - hunger) + (100 - prospective food consumption)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, M.D. PhD, Study Director — Steno Diabetes Center Copenhagen; Henriette H Nerild, M.D., Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided